CLINICAL TRIAL: NCT00506987
Title: Study of the Efficacy and Safety of SCH 486757 in Subjects With Chronic Idiopathic Cough
Brief Title: Study of the Efficacy and Safety of SCH 486757 in Subjects With Chronic Cough (Study P04887)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P04887; SCH 486757
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — 8-(bis(2-chlorophenyl)methyl)-3-(2-pyrimidinyl)-8-azabicyclo(3.2.1)octan-3-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCH 486757 (Experimental)
  Interventions: Drug: SCH 486757
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Dose 1

INTERVENTIONS:
Drug: SCH 486757 — SCH 486757 2 x 50-mg capsule twice daily orally for 2 weeks followed by a 2-week washout period and 2 weeks of crossover treatment
  Arms: SCH 486757
Drug: Placebo Dose 1 — Matching placebo capsules twice daily orally for 2 weeks followed by a 2 week washout period and 2 weeks of crossover treatment
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, crossover, single center study of SCH 486757 in subjects with chronic cough. Subjects will be randomized to receive SCH 486757 or placebo for 14 days. After a 2-week washout period, subjects will be crossed over to the other treatment. The primary objective is to evaluate the effectiveness of SCH 486757 in reducing cough reflex sensitivity as determined by a challenge with capsaicin, an agent that induces cough.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18 to <65 years old, with a history of a dry cough for >6 months.
* By history, evaluation of gastroesophageal reflux disease was done and ruled out by a minimum of an 8-week trial of antacid therapy (with a proton-pump inhibitor [PPI] given twice daily) with no clinical response in cough.
* By history, if there are clinical signs and symptoms of postnasal drip, these signs and symptoms will have been treated with a combination of an antihistamine and decongestant for a minimum of 8 weeks with no clinical response in cough.
* By history, if there are clinical signs and symptoms of asthma, these signs and symptoms will have been treated with a combination of an inhaled steroid and a short-acting beta-agonist for a minimum of 8 weeks with no clinical response in cough.

Exclusion Criteria:

* Subjects with current evidence of clinically significant pulmonary (especially conditions that involve coughing), hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric, autoimmune, or other disease that precludes the subject's participation in the study. In particular, diabetics, uncontrolled hypertensives, and subjects with clinically significant cardiomyopathy, prostatic hypertrophy, glaucoma, seizure disorders, and psychiatric disorders are to be excluded from participation in this study.
* Subjects with asthma or chronic obstructive pulmonary disease who require chronic use of inhaled or systemic corticosteroids.
* Subjects receiving concurrent prohibited medications unless they observe the washout period prior to the baseline visit. These medications would include opioid- and non-opioid-containing cough suppressants and potent CYP3A inhibitors, such as ritonavir, ketoconazole, and clarithromycin. Subjects receiving ACE inhibitors or MAOIs will be excluded from the study.
* Subjects with a history of allergies to more than two classes of medications.
* Current smokers, ex-smokers who stopped smoking in the previous 6 months, or subjects with a cumulative smoking history >10 pack-years will be excluded. (Pack-years is a way to measure the amount a person has smoked over a long period of time. It is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked, eg, a 10 pack-year history is equal to smoking 1 pack per day for 10 years or 2 packs per day for 5 years, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cough reflex sensitivity as assessed by log10 C5 resulting from a capsaicin challenge. A capsaicin challenge will be performed on the first day (before dosing) and on the last day of each 2 week treatment period. | After 2 weeks of treatment.

SECONDARY OUTCOMES:
Change from baseline in hourly cough rate over 24 hours (using an automated cough counter). Baseline will be measured as the total no. of coughs on Day 1 of each treatment period and compared with the same value on the last day of each treatment period. | After 2 weeks of treatment.